CLINICAL TRIAL: NCT00532584
Title: Effect of Inhaled Steroids in Combination With a Long Acting Bronchodilator on Gene Expression in the Lungs of Healthy Smokers
Brief Title: Effect of Steroids on Gene Expression in the Healthy Smokers Lungs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not initiated due to funding.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0709009398
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; inhaled steroids; bronchodilator; gene expression; smoker's lungs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- treatment with inhaled beclomethasone (Experimental): The treatment with inhaled beclomethasone will be administered to Group A from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. QVAR will be purchased by the Department of Genetic Medicine. The dose will be 2 puffs twice a day for 7 days
  Interventions: Drug: Beclomethasone
- Control - healthy smokers (No Intervention): Group B will act as control and include healthy smokers who receive no treatment.
- control - healthy non-smokers (No Intervention): Group C will act as control and include healthy non-smokers who receive no treatment.

INTERVENTIONS:
Drug: Beclomethasone — The treatment with inhaled beclomethasone will be administered to Group A from Day 1 to Day 7 via a metered dose inhaler (QVAR 80 HFA) delivering 80 micrograms of beclomethasone per puff. QVAR will be purchased by the Department of Genetic Medicine. The dose will be 2 puffs twice a day for 7 days
  Arms: treatment with inhaled beclomethasone

SUMMARY:
Cigarette smoking is the main risk factor for chronic obstructive pulmonary disease (COPD). The cells lining the lung airways (epithelium) and the cells on the surface of the epithelium (alveolar macrophages) of healthy smokers develop characteristic gene expression changes that are different from that of nonsmokers. These gene expression changes include up- and down-regulation of genes in functional categories known to be relevant to the development of COPD. Administration of anti-inflammatory medications (inhaled steroids) in combination with long acting medications that open the airways (bronchodilators), are known to decrease the rate of acute exacerbations and improve the quality of life of individuals with COPD; however, the mechanisms underlying these beneficial effects of are poorly understood. This study will assess the effect of traditional therapy for COPD (inhaled corticosteroids, an anti-inflammatory medication, plus a bronchodilator, a medication that helps open the airways) on smoking-induced gene changes in airway epithelium and alveolar macrophages. Volunteer subjects will be evaluated by bronchoscopy to sample lung cells at 0, 7 and 14 days, with the therapy given at day 1 through day 7. The bronchoscopy aspects of this study will be covered by approved Weill-Cornell IRB protocol # 0005004439 (see below.)

To participate in this protocol, the research subject will first be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy", fulfilling the inclusion/exclusion criteria of that protocol. They will be invited to participate in this protocol only if they meet the additional inclusion/exclusion criteria of this protocol.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of inhaled beclomethasone (an inhaled corticosteroid) on the pattern of the lung airway epithelium and alveolar macrophages gene expression of healthy smokers. We hypothesize that the administration of beclomethasone will result in reversibility of some of the airway epithelium and alveolar macrophage gene expression changes induced by cigarette smoking.

Background. Chronic obstructive pulmonary disease (COPD), including chronic bronchitis and emphysema, occurs in 15 to 20% of individuals who smoke, and is a leading cause of disease and mortality in the US (1, 2). Cigarette smoking is found to be the cause of approximately 90% of the cases of COPD in the US (1, 2). The human lung airway epithelium receives the initial brunt of cigarette smoking, and the airway epithelium and alveolar macrophages play a central role in the development of COPD (3-6). Asymptomatic healthy smokers have increased rate of cell proliferation in the airway epithelium consistent with the concept that the airway epithelium of smokers undergoes molecular changes that precede the development of COPD (7). Similarly, smoking increases the number and activates the alveolar macrophages present in the alveoli of human lung leading to the release of various mediators involved in the pathogenesis of COPD (4, 6, 8, 9).

Assessment of human lung airway epithelium and alveolar macrophages gene expression of healthy smokers compared to healthy non-smoking individuals demonstrate that the epithelium of the large and the small airways and the alveolar macrophages up- and down-regulate a variety of genes relevant to the pathogenesis of COPD (10-15). The differential gene expression in the epithelium of smokers compared to nonsmokers comprises genes in various functions, including genes involved in inflammation, cell repair, cell differentiation, cell death, detoxification, and cell signaling. While the airway epithelium is target for the stress of cigarette smoking, alveolar macrophages (the pulmonary representative of the bone marrow-derived mononuclear phagocyte system) are activated by smoking, and release a variety of mediators that can injure the fragile lung structure (4, 6, 16). Thus, while the airway epithelium is injured by smoking, the alveolar macrophages contribute to the smoking-induced injury. Many studies in vitro and in vivo in animals and in humans demonstrate the role of the airway epithelium and alveolar macrophages in the development of COPD with the release of various pro-inflammatory mediators, and mediators involved in cell apoptosis, proteolysis, airway remodeling and obstruction contributing to the characteristic findings of inflammation and obstruction observed in the airways of individuals with COPD (3-9, 17, 18).

Beclomethasone is one of the medications that when administered by inhalation to individuals with moderate to severe COPD results in reduction of hospitalization by approximately 30%, increased quality of life, and a decreased in the reduction of lung function (19, 20). Interestingly, beclomethasone is one of the medications that when administered by inhalation following hospitalization with acute exacerbation to individuals with COPD, results in a lower re-hospitalization rate. The mechanisms by which inhaled steroids result in clinical improvement and increased quality of life in individuals with moderate to severe COPD and following acute exacerbations are poorly understood (19-24).

ELIGIBILITY:
Inclusion Criteria:

Group A and B

* All study individual should be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
* All study subjects should be able to provide informed consent
* Current smokers with 15-to 40 pack-year history
* All study individuals should be healthy as per protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"

Group C

* All study individual should be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"
* All study subjects should be able to provide informed consent
* All study individual should be healthy as per protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy"

Exclusion Criteria:

Group A and B

* Smokers intending to quit smoking in the next 14 days.
* Individuals already receiving any lung related inhalers
* Females who are pregnant or nursing

Group C

Exclusion Criteria:

* Non-smokers who intend to start smoking in the next 14 days
* Individuals already receiving any lung related inhalers
* Females who are pregnant or nursing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Microarray chips are scanned and analyzed using Affymatrix Microarray suite version 5 (MAS5). Using GeneSpring software the data is normalized and differential expression is determined using alveolar macrophages. | Day 7 and Day 14 following initiation of therapy compared to baseline values obtained on screening

SECONDARY OUTCOMES:
St. George Respiratory questionnaire | To be completed on Screening Day

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Tilley, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided